CLINICAL TRIAL: NCT04555434
Title: Effects of Probiotics (P. Pentosaceus, L. Lactis or L. Helveticus) in Patients With Nonalcoholic Hepatitis
Brief Title: Effects of Probiotics (P. Pentosaceus, L. Lactis or L. Helveticus) in NASH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chuncheon Sacred Heart Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: PRO-NASH
Record Dates: First submitted 2020-07-01; First posted 2020-09-18 (Actual); Last update posted 2020-09-18 (Actual); Status verified 2020-07

CONDITIONS: Non-Alcoholic Fatty Liver Disease
Keywords: Probiotics; Liver disease; Gut microbiota
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Liver Diseases | interventions — Probiotics; Cellulose

STUDY DESIGN:
Intervention Model Description: Evaluates the effect of probiotic improvement on non-alcoholic fatty liver disease in patients diagnosed with non-alcoholic fatty liver disease.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotics group (Experimental): The selected test subjects were randomly assigned to test group 1, test group 2, test group 3, or control group according to the order registered at visit 2 (week 0) after a 2-week run-in period, and for 8 weeks, the study drug or study After taking the treaty, analyze the results of the observations.
  Interventions: Dietary Supplement: Probiotics
- Placebo group (Placebo Comparator): The selected test subjects were randomly assigned to test group 1, test group 2, test group 3, or control group according to the order registered at visit 2 (week 0) after a 2-week run-in period, and for 8 weeks, the study drug or study After taking the treaty, analyze the results of the observations.
  Interventions: Dietary Supplement: Probiotics

INTERVENTIONS:
Dietary Supplement: Probiotics — * Experimental group Main ingredients: P. pentosaceus KID7, L. lactis CKDB001 or L. helveticus CKDB001 (containing 9 × 10^9 CFU / day)
  * Control group Main ingredient: Crystalline cellulose
  Other Names: Cellulose (Placebo)

SUMMARY:
A study for evaluating the improvement effect of non-alcoholic steatohepatitis (NASH) of probiotics

DETAILED DESCRIPTION:
Non-alcoholic fatty liver disease progresses to fatty liver, hepatitis, cirrhosis, and liver cancer, resulting in a high mortality rate. The prevalence of non-alcoholic fatty liver disease at home and abroad is a major social and economic burden. However, there is no cure for non-alcoholic fatty liver disease. Recently, intestinal axis theory related to the development of chronic liver disease and microbial community has emerged. Intake of probiotics is known to play a role in regulating gut microflora. Improvement of non-alcoholic fatty liver disease can be expected through administration of probiotics.

ELIGIBILITY:
Inclusion Criteria:

1. Those who agreed to participate in this study and signed a written consent
2. Adult men and women over 20
3. Patients diagnosed with non-alcoholic fatty liver

   ※ Exclusion criteria for alcoholic liver disease
   * Those who have an alcoholic drinking ability of at least 60g per day for at least one year before visiting (30g for women)
   * 1 bottle of shochu 360 ml * 20% = 72 g, 1 bottle of beer 500 ml (330 ml for commercial use) * 5% = 25 (16.5 g)
4. Patients with higher liver numbers than normal ※ Adult normal liver level range by enzyme

   * AST, ALT: 40 or less
   * ALP: 20-130
   * GOT: 0-30, GPT: 0-38
   * GGT: 10-62 (male), 7-35 (female)

Exclusion Criteria:

1. Those who have consumed probiotics (lactic acid bacteria, etc.), prebiotics (dietary fiber, fructooligosaccharide, etc.), new biotics, fermented milk, etc. within the past month.
2. Those who have continuously taken antibiotics within the last 2 months or who are likely to take them during the study period
3. Those who have continuously consumed medicines or health functional foods that affect liver function within the past month.
4. Those who have participated in other clinical trials within the past 1 month (but not applicable to medical device clinical trials)
5. If you have any of the following

   * Alcoholic liver disease, hereditary metabolic disease, autoimmune hepatitis
   * systemic inflammatory disease or immune disease
   * Hepatocellular carcinoma
   * Uncontrolled cardiopulmonary disease
   * Other serious systemic disorders in the heart, lungs, blood, and endocrine system
6. A person with a history of malignancy diagnosis within the last 5 years
7. Pregnant or lactating women
8. Persons who have hypersensitivity to the test drug / placebo or components contained in the test drug / placebo or have severe allergic reactions
9. Those who are not suitable for the clinical trial because the investigator judges

Ages: 21 Years to 62 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-09-11 (Estimated); Study Completion 2020-09-11 (Estimated)

PRIMARY OUTCOMES:
Demographic characteristics | 1 week
  The gender, date of birth, age, menstruation, and amenorrhea, FAMILY HISTORY
Primary Outcomes; Liver Function Test | Baseline of AST, ALT, rGT, CHOL, and ALP at first week.
  Primary outcomes of liver function enzyme level (AST, ALT, rGT, CHOL, ALP)[IU/L]
Gut-Microbiome Composition | Change from Baseline of fecal microbiome at 8 months
  Change of the species and proportions of the gut microbiome. Proportion of phyrum level Composition of F/B ratio
Computed Tomography | Change from Baseline of CT image at 8 months
  change of the Abdominal ultrasonography or Computed Tomography(CT): Upper abdominal ultrasound or CT to determine the degree of fatty liver disease
  ② Fibroscan: Objectively and quantitatively grasp the degree of liver fibrosis by measuring the degree of firmness (elasticity) of the liver
change of BMI | Change from Baseline BMI and weight at 6 months
  Compare the body mass index. BMI=Body Weight/(Height)^2
Secondary Outcomes; Liver Function Test | Change from Baseline of AST, ALT, rGT, CHOL, and ALP at 8 months
  Secondary outcomes of liver function enzyme level (AST, ALT, rGT, CHOL, ALP)[IU/L]

CONTACTS AND LOCATIONS:
Locations (1):
- Hallym University Chuncheon Sacred Heart Hospital, Chuncheon, Gangwon-do, South Korea

REFERENCES:
- [Derived] Won SM, Joung H, Park IG, Han SH, Ham YL, Han JS, Kwon Y, Kim DJ, Suk KT. The effects of next generation probiotics on metabolic dysfunction-associated steatotic liver disease: a parallel, double-blind, randomized, placebo-controlled trial. J Transl Med. 2025 Dec 9;24(1):61. doi: 10.1186/s12967-025-07478-z. PMID 41366779